CLINICAL TRIAL: NCT05290142
Title: A Pre-and-post Study With a Nested Randomised Controlled Trial of Coach Versus Self-guided Digital Training in a Youth-focused Problem-solving Intervention
Brief Title: Pre-and-post Study With a Nested Randomized Trial of Digital Training to Teach Problem-solving Counselling in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sangath (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: VP_2015_017; 106919/Z/15/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-05

CONDITIONS: Depression, Anxiety
Keywords: digital training; mental health intervention; adolescent mental health; non-specialists
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Interventional Study Model: Digital training intervention: delivered to all participants (pre-and-post comparison) Additional coaching intervention: two-arm, individually randomized controlled trial with parallel assignment
Who Masked: Participant, Investigator
Masking Description: Double (Investigator, Outcomes Assessor). Participants will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Guided Digital Training (DT) (Active Comparator): Participants will be enrolled in a digital training course that addresses non-specific counselling skills and skills specific to an evidence-based problem-solving intervention. The course will be available online on a smartphone app as well as a website that can be accessed through an internet-enabled device.
  Participants will also have an option to message a centralized helpline for assistance with accessing and navigating the digital interface.
  Interventions: Other: Self-Guided Digital Training
- Digital Training with Coaching (DT-C) (Experimental): In addition to receiving the same digital training resources as the DT group, participants in DT-C will receive weekly individualized telephone calls from a coach who will motivate them and troubleshoot towards course completion. Participants will also be able to send text messages to coaches.
  Interventions: Other: Digital Training with Coaching (DT-C)

INTERVENTIONS:
Other: Digital Training with Coaching (DT-C) — An identical digital training course and helpline will be available for the participants in this group. In addition to receiving the same digital training resources as the DT group, participants in DT-C will receive weekly individualized telephone calls from a coach who will motivate them and troubleshoot towards course completion. The focus will be on clarifying learning objectives and redirecting participants to relevant materials rather than providing new learning opportunities. Participants will also be able to send text messages to coaches with queries related to course content, progress and technical difficulties. Coaches will reply to participants' messages within one working day and send reminders about upcoming telephone sessions, as well as prompts if the participant has not logged into the course for 3 consecutive days.
  Arms: Digital Training with Coaching (DT-C)
Other: Self-Guided Digital Training — Participants will be enrolled in a digital training course that addresses non-specific counselling skills and skills specific to an evidence-based problem-solving intervention. The course will be available offline and online on a smartphone app (called 'Sangath Training') as well as a website (https://training.sangath.in/login/index.php) that can be accessed through an internet-enabled device. The training will be delivered through didactic lectures, role-play demonstrations, and recommended readings spread across 16 modules. Participants will be provided with automated feedback on their learning through self-assessment quizzes after each module. Modules will be available sequentially and unlocked after accessing all content in the preceding module, over a period of 4 weeks. Technical helpline: Participants will also have an option to message a centralized helpline for assistance with accessing and navigating the digital interface.
  Arms: Self-Guided Digital Training (DT)

SUMMARY:
This study is part of a Wellcome Trust-funded research program in India called PRIDE (PRemIum for aDolEscents, 2016-2022) led by Principal Investigator Prof. Vikram Patel (Harvard Medical School). The goal of PRIDE is to establish a suite of scalable psychosocial interventions for common adolescent mental health problems in India.

Following on from earlier studies to develop and evaluate the various PRIDE interventions in school settings, the current study aims to generate evidence on methods to support implementation. We will undertake a pre-and-post study design with a nested randomized controlled trial with the specific aims to:

1. Evaluate the effects of digital training on non-specialists' competency to deliver an evidence-based problem-solving intervention for common adolescent mental health problems
2. Evaluate the incremental effect of digital training with coaching (DT-C) in comparison with self-guided digital training (DT) on non-specialists' competency to deliver an evidence-based problem-solving intervention for common adolescent mental health problems
3. Evaluate the processes affecting the implementation of training interventions in both arms

DETAILED DESCRIPTION:
PRIDE has been implemented in India to address the scarcity of evidence- based interventions for common adolescent mental health problems nationally and in low-resource settings more widely (Michelson et al., 2020). The goal is to develop and evaluate a suite of scalable, transdiagnostic psychological interventions (i.e., suitable for a variety of mental health presentations) that can be delivered by non-specialist ('lay') counsellors in resource-poor school settings.

There is a major knowledge gap concerning how to build capacity outside of specialist health settings and how to motivate and support non-specialists through structured capacity building activities in absence of adequate specialist trainers.

Hence, the aim of the current study is to evaluate the effectiveness of a digital training for non-specialists to improve their competency in delivering an evidence-based adolescent mental health intervention.

SIGNIFICANCE:

The health care system in India faces a number of key challenges: (1) poor quality and inadequately resourced primary health care; (2) low numbers and unequally distributed skilled human resources; (3) a large, unregulated, private sector; (4) low public spending on health leading to high levels of out of pocket expenditure; (5) fragmented health information systems; (6) irrational use and spiralling costs of drugs and technology; and (7) weak governance and accountability.

The current study will address the dearth of evidence on workforce development strategies necessary to scale-up evidence-based adolescent mental health interventions in low-resource settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Associated with one of the partner organizations/institutes
* Access to an internet-enabled smartphone or computer device
* Provides consent to participate

Exclusion Criteria:

* Prior practice-based education and/or training in psychotherapy or mental health interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Knowledge quiz | Change from Baseline Knowledge-based Competency at 6 weeks post randomisation
  The primary outcome is a knowledge-based competency measure that incorporates an 17-item multiple-choice quiz (MCQ), with questions related to case-based vignettes that will be administered through the REDCap platform. Parallel forms of the quiz will be used at baseline and endline assessments, the sequencing of which will be determined at random. The assessment format and topic domains have been informed by previous research on competency assessments for nonspecialists (Asher et al., 2021; Ottman, Kohrt, Pedersen & Schafer, 2020; Pedersen et al., 2021; Kohrt et al. 2015a; Kohrt et al. 2015b, Kohrt et al. 2020). The measure includes questions related to psychotherapies generally as well as specific problem-solving competencies.). Prior to unblinding the dataset, we will carry out a psychometric analysis of MCQ item scores across the entire sample. Poorly performing items may be removed and the primary outcome analysis will be conducted using retained items.

SECONDARY OUTCOMES:
MUSIC | 6 weeks post randomisation
  This will be assessed post-training only. We will use a 26-item questionnaire adapted from MUSIC (eMpowerment, Usefulness, Success, Interest, Caring), an established measure of satisfaction with educational programs that has previously been used in the study setting (Jones, 2017). Items on the questionnaire cover the feasibility, acceptability, adoption and appropriateness of the training program. These are rated on 6 point likert scale ranging from Strongly Agree to Strongly Disagree. The purpose is to identify strengths and weaknesses related to course content that may influence participants' engagement and thus to inform improvements.

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Patel, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (9):
- India (9):
  - Acharya Institue, Bangalore, Karnataka
  - Maniben Nanavati Women's College, Mumbai, Maharashtra
  - Ballygunj Society for Children in Pain, Mumbai, Maharashtra
  - Al-Falah University, New Delhi, National Capital Territory of Delhi
  - Agragami India, New Delhi, National Capital Territory of Delhi
  - Youth for Mental Health, New Delhi, National Capital Territory of Delhi
  - Christ University, Ghaziabad, Uttar Pradesh
  - YP Foundation, Noida, Uttar Pradesh
  - World Health Partners, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Plan to Share IPD: Anonymised participant data, data dictionary and case report forms will be made available 12 months after study completion. Data will be shared after approval by the corresponding author, following a reasonable submitted request. The study protocol and statistical analysis plan are publicly available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after study completion
Access Criteria: Access to data will be granted to researchers after review of requests by the PI and in accordance with the guidelines of sponsors, collaborators and the study funder.

REFERENCES:
- [Background] Michelson D, Malik K, Parikh R, Weiss HA, Doyle AM, Bhat B, Sahu R, Chilhate B, Mathur S, Krishna M, Sharma R, Sudhir P, King M, Cuijpers P, Chorpita B, Fairburn CG, Patel V. Effectiveness of a brief lay counsellor-delivered, problem-solving intervention for adolescent mental health problems in urban, low-income schools in India: a randomised controlled trial. Lancet Child Adolesc Health. 2020 Aug;4(8):571-582. doi: 10.1016/S2352-4642(20)30173-5. Epub 2020 Jun 23. PMID 32585185
- [Background] Asher L, Birhane R, Teferra S, Milkias B, Worku B, Habtamu A, Kohrt BA, Hanlon C. "Like a doctor, like a brother": Achieving competence amongst lay health workers delivering community-based rehabilitation for people with schizophrenia in Ethiopia. PLoS One. 2021 Feb 25;16(2):e0246158. doi: 10.1371/journal.pone.0246158. eCollection 2021. PMID 33630893
- [Background] Ottman KE, Kohrt BA, Pedersen GA, Schafer A. Use of role plays to assess therapist competency and its association with client outcomes in psychological interventions: A scoping review and competency research agenda. Behav Res Ther. 2020 Jul;130:103531. doi: 10.1016/j.brat.2019.103531. Epub 2019 Dec 14. PMID 31902517
- [Background] Pedersen, G. A., Gebrekristos, F., Eloul, L., Golden, S., Hemmo, M., Akhtar, A., ... & Kohrt, B. A. (2021). Development of a Tool to Assess Competencies of Problem Management Plus Facilitators Using Observed Standardised Role Plays: The EQUIP Competency Rating Scale for Problem Management Plus. Intervention, 19(1), 107.
- [Background] Kohrt BA, Jordans MJ, Rai S, Shrestha P, Luitel NP, Ramaiya MK, Singla DR, Patel V. Therapist competence in global mental health: Development of the ENhancing Assessment of Common Therapeutic factors (ENACT) rating scale. Behav Res Ther. 2015 Jun;69:11-21. doi: 10.1016/j.brat.2015.03.009. Epub 2015 Mar 24. PMID 25847276
- [Background] Kohrt BA, Ramaiya MK, Rai S, Bhardwaj A, Jordans MJD. Development of a scoring system for non-specialist ratings of clinical competence in global mental health: a qualitative process evaluation of the Enhancing Assessment of Common Therapeutic Factors (ENACT) scale. Glob Ment Health (Camb). 2015;2:e23. doi: 10.1017/gmh.2015.21. Epub 2015 Dec 9. PMID 28593049
- [Background] Kohrt BA, Schafer A, Willhoite A, Van't Hof E, Pedersen GA, Watts S, Ottman K, Carswell K, van Ommeren M. Ensuring Quality in Psychological Support (WHO EQUIP): developing a competent global workforce. World Psychiatry. 2020 Feb;19(1):115-116. doi: 10.1002/wps.20704. No abstract available. PMID 31922690
- [Background] Jones, B. D., Li, M., & Cruz, J. M. (2017). A cross-cultural validation of the MUSIC® Model of Academic Motivation Inventory: Evidence from Chinese-and Spanish-speaking university students. International Journal of Educational Psychology, 6(1), 25-44.
- [Derived] Mathur S, Weiss HA, Neuman M, Field AP, Leurent B, Shetty T, J JE, Nair P, Mathews R, Malik K, Michelson D, Patel V. Coach-Supported Versus Self-guided Digital Training Course for a Problem-solving Psychological Intervention for Nonspecialists: Protocol for a Pre-Post Nested Randomized Controlled Trial. JMIR Res Protoc. 2023 Jun 13;12:e41981. doi: 10.2196/41981. PMID 37310781

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT05290142/SAP_000.pdf